CLINICAL TRIAL: NCT05580237
Title: Pressure Gradient vs. Flow Relationships in Patients With Symptomatic Valvular Aortic Stenosis - a Comparison Between High- and Low Gradient Subtypes
Brief Title: Pressure Gradient vs. Flow Relationships in Patients With Symptomatic Valvular Aortic Stenosis
Acronym: PREFLOW
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Henrik Vase, Staff Specialist, MD, PhD, Aarhus University Hospital Skejby
Other Study IDs: 1-10-72-71-19
Record Dates: First submitted 2022-05-10; First posted 2022-10-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe aortic valve stenosis
  Interventions: Procedure: Simultaneous right and left heart catheterization

INTERVENTIONS:
Procedure: Simultaneous right and left heart catheterization — Pressure recordings across the aortic valve with simultaneous flow measurements by right heart catheterization, during rest and during supine exercise.

SUMMARY:
The objective of the present study is to investigate to hemodynamic profile at rest and during peak exercise of patients with suspected severe aortic stenosis and to compare flow- and pressure changes between high gradient patients and low gradient patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected severe AS scheduled for evaluation for aortic valve intervention:
* LVEF > 50 %
* AVA < 1.0 cm2
* Symptomatic - at least equivalent to NYHA functional class II

Exclusion Criteria:

* Congenital heart disease
* Severe coronary artery disease (main stem, proximal LAD or 3 vessel disease)
* Moderate or severe aortic valve regurgitation
* Moderate or severe mitral valve regurgitation or stenosis
* Moderate or severe pulmonary valve regurgitation or stenosis
* Moderate or severe tricuspid valve regurgitation or stenosis
* Severe pulmonary hypertension (tricuspid valve pressure gradient of 60 mmHg)
* Right ventricular dysfunction (TAPSE < 17 mm)
* Restrictive cardiomyopathy or cardiac amyloidosis
* Constrictive pericarditis
* Inability to perform supine bicycle exercise

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected severe AS scheduled for evaluation for aortic valve intervention
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pressure and flow relationships across the aortic valve during rest and during supine exercise | 2 hours
  Pressure drop across the aortic valve measured invasively. Flow across the valve estimated by right heart catheterization in the absence of aortic valve regurgitation.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Vase, MD, PhD, Principal Investigator — Department of Cardiology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark